CLINICAL TRIAL: NCT03632772
Title: Comparative Study of Solifenacin and Mirabegron in Treatment of Overactive Bladder Symptoms in Men After Transurethral Resection of the Prostate - A Randomized Prospective Study
Brief Title: Comparison of Solifenacin and Mirabegron in Treatment of Overactive Bladder Symptoms in Men After TURP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Buddhist Tzu Chi General Hospital (Other)
Responsible Party: Principal Investigator, Hann-Chorng Kuo, Chairman and Professor, Department of Urology, Buddhist Tzu Chi General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TCGH107-115-A
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2018-08-24 (Actual); Status verified 2018-08

CONDITIONS: Overactive Bladder Syndrome
Keywords: Overactive bladder; Transurethral Resection of the Prostate; Pharmacotherapy; Mirabegron; Solifenacin
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate; mirabegron

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Solifenacin 5 mg for 4 weeks (Experimental): Solifenacin 5 mg once-daily for 4 weeks.
  Interventions: Drug: Solifenacin 5Mg
- Mirabegron 50 mg for 4 weeks (Experimental): Mirabegron 50 mg once-daily for 4 weeks.
  Interventions: Drug: Mirabegron 50 MG
- Control: non treatment (No Intervention): Control: non treatment.

INTERVENTIONS:
Drug: Solifenacin 5Mg — We compared the safety and therapeutic efficacy between Solifenacin and Mirabegron in men with benign prostate hyperplasia and having overactive bladder symptoms immediately after Transurethral Resection of the Prostate.
  Other Names: Vesicare
  Arms: Solifenacin 5 mg for 4 weeks
Drug: Mirabegron 50 MG — We compared the safety and therapeutic efficacy between Solifenacin and Mirabegron in men with benign prostate hyperplasia and having overactive bladder symptoms immediately after Transurethral Resection of the Prostate.
  Other Names: Betmiga
  Arms: Mirabegron 50 mg for 4 weeks

SUMMARY:
Urinary frequency urgency and urgency urinary incontinence (UUI) are commonly encountered in patients after transurethral prostatectomy (TURP) or transurethral incision of the prostate (TUIP). Antimuscarinics has been widely used to treat OAB and around 70% of patients can improve symptoms after treatment. Beta-3 adrenoceptor agonist (mirabegron) can also decrease DO and improve OAB symptoms. Combination treatment of solifenacin 5mg plus mirabegron 25 or 50mg was more effective than mirabegron 50mg alone, but with more anticholinergic side effects. However, there has been no clinical trial to compare which drug provides more benefit to decrease the OAB symptom severity immediately after TURP. This study tries to compare the safety and therapeutic efficacy between solifenacin and mirabegron in men with BPH and having OAB symptoms immediately after TURP.

This study was designed as a prospective, randomized trial to compare the safety and efficacy of OAB medication on the decrease of overactive bladder symptoms score (OABSS) and urgency severity score (USS) between solifenacin 5mg QD and mirabegron 50mg QD in men with BPH undergoing TURP. A total of 130 male patients with BPH and undergo TURP or TUIP will be enrolled. The primary end point is the change of USS from baseline to 4 weeks after catheter removal and starting OAB medication. Secondary end-points include the changes of OABSS, frequency episodes, urgency episodes, UUI episodes in the 3-day voiding diary, maximum flow rate (Qmax), voided volume and PVR, International Prostate Symptom Score (IPSS) and quality of life index (QoL-I) from baseline to 2 weeks and 4 weeks.

We expect that patients receiving solifenacin and mirabegron might have similar therapeutic effects on decrease of USS, but patients who received mirabegron might have less adverse events such as dry mouth or difficulty in urination.

DETAILED DESCRIPTION:
Introduction:

Urinary frequency urgency and urgency urinary incontinence (UUI) are commonly encountered in patients after transurethral prostatectomy (TURP) or transurethral incision of the prostate (TUIP). [1] Patients usually bother by these overactive bladder (OAB) symptoms. The causes of postprostatectomy OAB might be detrusor overactivity (DO) before TURP, increase afferent input due to acute inflammation after TURP, or a weak urethral sphincter which cannot hold urine at the bladder capacity. Antimuscarinics and beta-3 adrenoceptor agonist are two different classes of medication for OAB. [2] Antimuscarinics has been widely used to treat OAB and around 70% of patients can improve symptoms after treatment. Beta-3 adrenoceptor agonist (mirabegron) can also decrease DO and improve OAB symptoms. Combination treatment of solifenacin 5mg plus mirabegron 25 or 50mg was more effective than mirabegron 50mg alone, but with more anticholinergic side effects. [3] However, antimuscarnics might decrease detrusor contractility and result in increase of postvoid residual (PVR) volume. Current clinical studies reveal that mirabegron does not impair detrusor contractility or increase PVR. [4] Under this consideration, mirabegron has been widely used to treat male lower urinary tract symptoms (LUTS) due to benign prostate hyperplasia (BPH). [5] However, there has been no clinical trial to compare which drug provides more benefit to decrease the OAB symptom severity immediately after TURP. This study tries to compare the safety and therapeutic efficacy between solifenacin and mirabegron in men with BPH and having OAB symptoms immediately after TURP.

Material and methods:

Objectives and Endpoints: This study was designed as a prospective, randomized trial to compare the safety and efficacy of OAB medication on the decrease of overactive bladder symptoms score (OABSS) and urgency severity score (USS) between solifenacin 5mg QD and mirabegron 50mg QD in men with BPH undergoing TURP.

Randomization: Permuted block randomization method will be applied to generate randomization codes. Each randomization number will be assigned to individual patient according to the time-sequence for screened patient become eligible.

Expected Results:

Patients receiving solifenacin and mirabegron might have similar therapeutic effects on decrease of USS, but patients who received mirabegron might have less adverse events such as dry mouth or difficulty in urination.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients with BPH and undergo TURP or TUIP.
2. Patients void smoothly after catheter removal.
3. No active urinary tract infection.
4. No gross hematuria or blood clot obstruction.
5. Patient or his care giver can complete voiding diary and report symptoms.

Exclusion Criteria:

1. Patients have overt neurological diseases such as cerebrovascular disease, senile dementia or spinal cord injury.
2. Patients have severe medical disease and completely immobile.
3. Patients have PVR larger than 150ml.
4. Patients do not have OAB after TURP.

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients with benign prostate hyperplasia (BPH) and undergo transurethral prostatectomy (TURP) or transurethral incision of the prostate (TUIP).
Enrollment: 130 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-07-31 (Estimated); Study Completion 2019-07-31 (Estimated)

PRIMARY OUTCOMES:
Urgency Severity Scale (USS) | from baseline to 4 weeks
  The change of USS from baseline to 4 weeks after catheter removal and starting OAB medication.

SECONDARY OUTCOMES:
Overactive Bladder Symptom Score (OABSS) | from baseline to 2 weeks and 4 weeks.
  The changes of OABSS
frequency episodes, urgency episodes, urgency urinary incontinence (UUI) episodes in the 3-day voiding diary | from baseline to 2 weeks and 4 weeks.
  The changes of frequency episodes, urgency episodes, urgency urinary incontinence (UUI) episodes in the 3-day voiding diary
maximum flow rate (Qmax) | from baseline to 2 weeks and 4 weeks.
  The changes of maximum flow rate (Qmax)
voided volume (Vol) | from baseline to 2 weeks and 4 weeks.
  The changes of voided volume (Vol)
Postvoid residual volume (PVR) | from baseline to 2 weeks and 4 weeks.
  The changes of Postvoid residual volume (PVR)
International Prostate Symptom Score (IPSS) | from baseline to 2 weeks and 4 weeks.
  The changes of International Prostate Symptom Score (IPSS)
quality of life index (QoL-I) | from baseline to 2 weeks and 4 weeks.
  The changes of quality of life index (QoL-I)

CONTACTS AND LOCATIONS:
Overall Officials: Hann-Chorng Kuo, M.D., Principal Investigator — Department of Urology, Buddhist Tzu Chi General Hospital, Hualien
Locations (1):
- Buddhist Tzu Chi General Hospital, Hualien City, Taiwan

IPD SHARING:
Plan to Share IPD: No
IPD was not planned to share.

REFERENCES:
- [Background] Seki N, Yuki K, Takei M, Yamaguchi A, Naito S. Analysis of the prognostic factors for overactive bladder symptoms following surgical treatment in patients with benign prostatic obstruction. Neurourol Urodyn. 2009;28(3):197-201. doi: 10.1002/nau.20619. PMID 18973143
- [Background] Yamada S, Ito Y, Nishijima S, Kadekawa K, Sugaya K. Basic and clinical aspects of antimuscarinic agents used to treat overactive bladder. Pharmacol Ther. 2018 Sep;189:130-148. doi: 10.1016/j.pharmthera.2018.04.010. Epub 2018 Apr 27. PMID 29709423
- [Background] Kelleher C, Hakimi Z, Zur R, Siddiqui E, Maman K, Aballea S, Nazir J, Chapple C. Efficacy and Tolerability of Mirabegron Compared with Antimuscarinic Monotherapy or Combination Therapies for Overactive Bladder: A Systematic Review and Network Meta-analysis. Eur Urol. 2018 Sep;74(3):324-333. doi: 10.1016/j.eururo.2018.03.020. Epub 2018 Apr 23. PMID 29699858
- [Background] Wada N, Iuchi H, Kita M, Hashizume K, Matsumoto S, Kakizaki H. Urodynamic Efficacy and Safety of Mirabegron Add-on Treatment with Tamsulosin for Japanese Male Patients with Overactive Bladder. Low Urin Tract Symptoms. 2016 Sep;8(3):171-6. doi: 10.1111/luts.12091. Epub 2015 Feb 17. PMID 27619782
- [Background] Nitti VW, Rosenberg S, Mitcheson DH, He W, Fakhoury A, Martin NE. Urodynamics and safety of the beta(3)-adrenoceptor agonist mirabegron in males with lower urinary tract symptoms and bladder outlet obstruction. J Urol. 2013 Oct;190(4):1320-7. doi: 10.1016/j.juro.2013.05.062. Epub 2013 May 30. PMID 23727415
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401